CLINICAL TRIAL: NCT02949479
Title: Dissociative Experience During the Offence in Sex Offenders : Clinical and Prognosis Correlates
Brief Title: Dissociation Investigation Study in Sex Offenders
Acronym: DISSO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: STUDY INVESTIGATORS HAVE LEFT THE INSTITUTION, THE DEPARTMENT NO LONGER HAS TIME TO INCLUDE
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-A01019-42
Record Dates: First submitted 2016-10-05; First posted 2016-10-31 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2021-12

CONDITIONS: Sex Offenses
Keywords: sex offenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dissociation Investigation in Sex Offenders (Other): The study will be proposed to the subjects after their usual clinical evaluation in the center for sexual offence, and to extend this evaluation by a specific focus on childhood abuse and neglect, trauma and dissociative history
  Interventions: Behavioral: Dissociation Investigation in Sex Offenders

INTERVENTIONS:
Behavioral: Dissociation Investigation in Sex Offenders — prevalence of a clinical dissociative state during the offence; secondary : correlations of dissociation with childhood abuse or neglect, with significant lifetime dissociative experience, post traumatic stress disorder or dissociative disorder (DSM-5), violence and sexual estimated risk using actuarial and professional structured judgement tools

SUMMARY:
Background: Adverse childhood experience have been described in sexual offenders but the link with the offence need to be further investigated. Investigators postulate that one of the clinical moderating factors could be dissociative experience, a consequence of these early adverse experiences reactivated during the offence. The purpose of the study is to estimate the prevalence of clinical dissociation during the offence in a male adult population referred to our center for a sexual offence and to explore its correlations with epidemiological and clinical data (personal, legal history, psychiatric comorbidities), clinical trauma and dissociation, prognosis estimates.

DETAILED DESCRIPTION:
The study will be proposed to the subjects after their usual clinical evaluation in the center for sexual offence and to extend this evaluation by a specific focus on childhood abuse and neglect trauma and dissociative history. After receiving complete information, the participants will sign the consent form and be referred to a unique on-site visit of approximately 2 hours long. During this visit, the participants will benefit from a psychiatric examination in search for clinical features of dissociation during the offence, lifetime dissociative experience, lifetime post-traumatic stress disorder; they will have to complete bioevaluation forms for dissociation (Dissociative Experience Scale) and childhood abuse and neglect (Childhood Experience of Care and Abuse). After this completion, they will benefit from a second part psychiatric examination, so as to complete the assessment and answer their questions if any.

ELIGIBILITY:
Inclusion Criteria:

* male subject referred to the center for having committed a sexual offense; social insurance affiliation

Exclusion Criteria:

* schizophrenia, mental retardation (IQ<70)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
point prevalence of clinical dissociation during the offence, assessed with the use of clinical examination (narrative and DSM-5 criteria) | 3 years
  the presence of a clinical dissociative state will be assessed retrospectively with the use of clinical examination.

SECONDARY OUTCOMES:
lifetime dissociation | 3 years
  lifetime dissociation measured by the Dissociative Experience Scale
childhood abuse or neglect | 3 years
  Childhood abuse ant Neglect assessed by the Childhood Experience of Care and Abuse (CECA)
psychiatric comorbidities | 3 years
  psychiatric comorbidities
prognosis issues | 3 years
  risk assessment tools scoring

CONTACTS AND LOCATIONS:
Overall Officials: Mouchet-Mages Sabine, PH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No